CLINICAL TRIAL: NCT05666505
Title: A Pilot Study to Assess Performance of a New Low-Cost Mobile Health Based Prototype Tympanometer
Brief Title: Evaluation of a New mHealth Tympanometer
Status: Completed | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 274552
Record Dates: First submitted 2022-12-13; First posted 2022-12-27 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss
Keywords: Rural; Screening; Tympanometer; Mobile health (mHealth); Otitis media; ML Algorithm
MeSH Terms: conditions — Hearing Loss; Otitis Media

STUDY DESIGN:
Intervention Model Description: Each participant will be first tested with prototype mHealth tympanometer, and then with a commercial tympanometer routinely used in clinical settings.
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- Tympanometer Comparison (Experimental): Both ears of each participant will be tested first with the prototype mHealth tympanometer followed by standard of care commercial tympanometer
  Interventions: Device: Prototype mHealth tympanometer; Device: Standard of care commercial tympanometer

INTERVENTIONS:
Device: Prototype mHealth tympanometer — The prototype mHealth tympanometer functions similarly to a commercial tympanometer. Tympanometers are designed to assess middle ear function by measuring changes in acoustic tone related to subtle movement of the tympanic membrane from an applied air pressure sweep. An audiologist will review the tympanogram tracings and classify results as Type A, B, or C.
Device: Standard of care commercial tympanometer — A commercial tympanometer routinely used as part of standard of care will be used as the comparison. Tympanometers are designed to assess middle ear function by measuring changes in acoustic tone related to subtle movement of the tympanic membrane from an applied air pressure sweep. An audiologist will review the tympanogram tracings and classify results as Type A, B, or C.

SUMMARY:
Children in rural and underserved communities experience a disproportionately high burden of infection-related hearing loss, which is often preventable with timely identification and follow-up care. A tympanometer is a device that evaluates the health of the middle ear but is often not used in screening programs due to barriers of high cost and need for trained professionals such as audiologists to use the device. To address these barriers, a low cost, lay friendly, mobile health (mHealth) prototype tympanometer has been developed. In addition, a machine learning (ML) algorithm has been designed to guide lay users to interpret tympanometer results, overcoming the need for audiologists. Broad implementation of the lay friendly tympanometer and ML algorithm will transform screening in areas where prevalence of infection-related hearing loss is high, and access to specialty care is limited.

In this study the prototype mHealth tympanometer will be evaluated against commercial tympanometry. It will be used by audiologists, an essential step before testing the performance of the device with lay users. Approximately 20 adult patients and 10 pediatric patients with various middle ear pathologies will be enrolled in the study, with the goal of obtaining 60 ears with data from both the prototype and commercial tympanometers. Audiologists will obtain tympanometry measurements on both ears of each participant and interpret the results, first with the prototype device and then with the commercial tympanometer that is typically used during a clinical evaluation. Tympanometry interpretation will include classification into one of 3 categories (Type A, B, or C). Agreement in results between the prototype and commercial devices will be assessed. Agreement between audiologist interpretations and the ML algorithm from the prototype mHealth tympanometer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Audiology Clinic for evaluation, where tympanometry is warranted for testing at the discretion of the audiologist
* Presence of various middle ear health states/pathologies that result in Type A, B, C tympanograms
* English-speaking

Exclusion Criteria:

* Children or adults with cognitive disabilities
* Unable to provide consent/assent
* Individuals who are unable to sit still
* Any other condition that in the opinion of the investigator, might interfere with the safe conduct of the study or place the participant at increased risk

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tympanometer Comparison
Started | 39
Completed | 38
Not Completed | 1
Not completed — Withdrawn due to caregiver consent obtained from non-legal guardian | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tympanometer Comparison
Number analyzed (Participants) | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 26
  More than one race | 0
  Unknown or Not Reported | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 11
  >=65 years | 11

OUTCOME MEASURES:

1. Primary Outcome: Classification Agreement Between Prototype mHealth Tympanometer and Commercial Tympanometer
Description: Audiologist will test each ear of the participant first with the prototype device, interpret the results into one of the three tympanogram categories (Type A/B/C) and record the results. The procedure will be repeated with a commercial device. Agreement between the two devices with respect to the classification categories will be assessed.
Time Frame: Same day as participant visit, up to 10 minutes
Population: The analytic sample is limited to ear-level results that produced a classification result of A/B/C for both devices. Ears were not included in the main analysis if data from one device or both devices were missing for that ear.
Measure: Number; unit: Percent Agreement
Units Other Than Participants: Ears
Arm/Group | Tympanometer Comparison
Number analyzed (Participants) | 33
Number analyzed (Ears) | 60
Percent Agreement | 93.33

2. Primary Outcome: Classification Agreement Between Audiologist and ML Algorithm Interpretations Using Prototype mHealth Tympanometer
Description: Tympanogram results collected using the prototype mHealth tympanometer will be run through the ML algorithm for classification into Type A/B/C. Agreement between the audiologist and the ML algorithm with respect to the classification categories will be assessed.
Time Frame: Same day as participant visit, up to 10 minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Kappa-statistic (Agreement)
Units Other Than Participants: Ears
Arm/Group | Tympanometer Comparison
Number analyzed (Participants) | 33
Number analyzed (Ears) | 60
Kappa-statistic (Agreement) | 0.81 [0.64 to 0.94]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed twice on the day of the audiology clinic visit, once after testing with mHealth tympanometer, and once upon completion of the audiology clinic visit.
Groups:
- Prototype mHealth Tympanometer; Standard of Care Commercial Tympanometer: Both ears of each participant will be tested first with the prototype mHealth tympanometer followed by standard of care commercial tympanometer
  Prototype mHealth tympanometer: The prototype mHealth tympanometer functions similarly to a commercial tympanometer. Tympanometers are designed to assess middle ear function by measuring changes in acoustic tone related to subtle movement of the tympanic membrane from an applied air pressure sweep. An audiologist will review the tympanogram tracings and classify results as Type A, B, or C.
  Standard of care commercial tympanometer: A commercial tympanometer routinely used as part of standard of care will be used as the comparison. Tympanometers are designed to assess middle ear function by measuring changes in acoustic tone related to subtle movement of the tympanic membrane from an applied air pressure sweep. An audiologist will review the tympanogram tracings and classify results as Type A, B, or C.
Arm/Group | Prototype mHealth Tympanometer | Standard of Care Commercial Tympanometer
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT05666505/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05666505/SAP_001.pdf